CLINICAL TRIAL: NCT01823965
Title: Intravitreal Injections of Ranibizumab With Deferred Laser Grid Laser Photocoagulation for Treatment of Diabetic Macular Edema With Visual Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLOMD
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

ARMS (1):
- ranibizumab (Experimental)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab

SUMMARY:
In the prospective monocentric open label trial patients with diabetic macular edema will be treated with intravitreal injections of ranibizumab given for 3 months then with laser grid at month 4. During follow-up a ranibizumab injection will be performed every 2 months in case of best-corrected visual acuity decreased more than 5 letters.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus (1 or2)
* decreased vision from Diabetic Macular Edema (study eye Best Corrected Visual Acuity<69 letters using E.T.D.R.S testing)
* macular edema

Exclusion Criteria:

* history of severe cardiac disease
* stroke within 12 months
* intraocular inflammation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of intravitreal injections of ranibizumab | 1 years

SECONDARY OUTCOMES:
best-corrected visual acuity | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France